CLINICAL TRIAL: NCT05852548
Title: Parent-Mediated Intervention for Families With Children With Autism and Feeding Challenges, Australia Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1428 Australia; A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison)
Record Dates: First submitted 2023-04-28; First posted 2023-05-10 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Parent-Child Relations; Meals; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: One group, pre, post-test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent-Mediated Intervention with ASD (Experimental): In-home intervention (1-2x/week) will occur with families with children with ASD, including direct intervention, parent coaching, and parent training.
  Interventions: Behavioral: Parent-Mediated Intervention

INTERVENTIONS:
Behavioral: Parent-Mediated Intervention — Children with ASD will participate in a 6-month parent-mediated intervention that will include direct intervention and parent education.

SUMMARY:
The goal is to expand a parent-mediated intervention for feeding challenges in children with autism with an Australian cohort, building on recent research and current successful models already being used. A parent-mediated intervention would primarily occur in the home environment, working with the parent to establish goals and implement the intervention based on their child's specific needs.

DETAILED DESCRIPTION:
Fifty families with a child with Autism spectrum disorder (ASD) will be asked to participate in 24 parent-mediated feeding intervention visits over approximately six-months. In addition, parents will be asked to participate in 6 to 8 parent training sessions in their home or by phone. Enrollment with two groups of families will be staggered to allow for any further adaptation and refinement of the protocol based on feedback from enrolled families.

All families will be asked to participate in an initial intake session that will include an overview of the intervention program, assessment of the intervention targets, parent interview, observation/videotape of a family mealtime, and complete standardized questionnaires on specific variables (e.g., developmental level, autism severity and sensory processing) that can influence feeding behaviors to further describe the population and explore potential confounding variables. The assessments and mealtime observation will assist in determining the child's current feeding challenges and targeted goals. Both parent and child will be asked to participate in a video-taped mealtime and free play time during a laboratory session at pre and post-intervention time points. During the laboratory session, both parent and child will be asked to wear a heart rate activity monitor that attached to their chest via a harness and an electrodermal skin conductance wrist band to allow for wireless physiological data collection. In addition, parents and children will also be requested to wear the heart rate activity monitor two times in their home environment during family mealtime. Hair samples will be taken from both the parent and the child to assess recent stress levels. Parents will collaborate in Goal Attainment Scaling to allow for a pre- and post-test comparison of child specific goals. In addition, feeding assessments as well as a parent stress measure, heart rate variability, and hair cortisol measurement will be used for a pre- and post-test comparison. Parents will participate in brief structured interviews before, one time during, and immediately following completion of the program to provide feedback on the intervention.

Intervention:

1. Parents will attend 8 group sessions that will be clustered in the first three quarters of the program focused on topics related to feeding challenges (e.g. goal setting, feeding development, parent-child interactions, sensory processing, behavior management, nutrition, the gastrointestinal system, and family mealtimes). Education sessions will be facilitated by the principal investigator and research team members.
2. Parents will receive 6-10 individual sessions with a feeding interventionist that will support targeted goal setting, problem solving and individual coaching and feedback through video review of parent-led intervention.
3. Parent-child dyads will receive 24 weekly sessions in the home that demonstrate modeling of intervention strategies and provide direct feedback of parent-led intervention. Parent satisfaction and burden will be assessed after each weekly session using a brief Likert scale questionnaire.
4. Parents will be asked to commit 10-15 hours per week in the home setting to directly support targeted feeding goals and related challenges such as sensory processing that may be a barrier to successful eating. Two trained individuals with experience working with children with ASD will be hired to support facilitation of the parent-mediated intervention. Several steps will be taken to train and supervise the interventionists. In addition, a minimum of 20% of their interactions will be video-taped reviewed by the principal investigator to monitor treatment fidelity.

Analysis:

Descriptive statistics will be used to describe the family and child characteristics as well as family satisfaction. Interview data from the parents will be audio recorded, transcribed verbatim and imported into Nvivo for data management and analysis support to inform future adaptations of the intervention program as well as beginning to unravel who the program may be most effective for and why. An analysis of variance (ANOVA) will be used to assess the pre- and post-intervention differences of the key variables of interest.

ELIGIBILITY:
Inclusion Criteria:

* Child with a confirmed diagnosis of ASD (ages 2-7 years)
* Parent reported feeding problems
* English Speaking

Exclusion Criteria:

* Any conditions co-morbid with ASD (e.g., fragile X)
* Significant visual, hearing or physical impairments
* Children who receive any non-oral nutritional supplementation (e.g. gastrostomy tubes)

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-06-24 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Change in Sensory Experiences Questionnaire (SEQ 3.0) | Pre/post measure through study completion, an average of 6 months
  Caregiver report instrument designed to characterize sensory features in children ages 2-12 years with ASD. This is a 105-item questionnaire, the scoring is based on the first 97: scored on a 5 point scale from 1 (almost never) to 5 (almost always). The remaining items are qualitative and provide context. Total possible range of scores is 97-485, higher scores indicate greater intensity of sensory behaviors.
Change in Goal Attainment Scaling (GAS) | Pre/Post measure through study completion, an average of 6 months
  Assesses the effectiveness of psycho-social interventions in the community setting in ASD. The total possible range of standardized T scores is 23.56 - 76.44, where a score of 50 means all goals were met and higher scores indicate goals were exceeded.
Change in Feeding and Eating in AutiSm Together Questionnaire | Pre/Post measure through study completion, an average of 6 months
  Measures feeding challenges across domains of sensory, behavior, oral motor, and gastrointestinal as well as how feeding challenges present in daily life and family routines. The total possible range of scores for each domain is from 32-160 with higher scores indicating increased feeding challenge.

SECONDARY OUTCOMES:
Change in the Caregiver Involvement Scale Score | Pre/Post intervention session measure through study completion, an average of 1 time per month (for up to 6 months)
  The Caregiver Involvement Scale is a 6-item instrument scored on a 5-point likert scale for a total possible range of scores from 6-30, where higher scores indicate increased caregiver comfort and involvement with the intervention.
Change in Parent effort scale | Pre/Post intervention session measure through study completion, an average of 1 time per month (for up to 6 months)
  Measures the amount of effort parents are applying to help their child complete daily activities. . 34-items about parental effort are scored on a 5-point likert scale from 1 (none) to 5 (too much to participate) for a total score of 34-170 where higher scores indicate increased parent effort.

CONTACTS AND LOCATIONS:
Overall Officials: Karla K Ausderau, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- La Trobe University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodak T, Piazza CC. Assessment and behavioral treatment of feeding and sleeping disorders in children with autism spectrum disorders. Child Adolesc Psychiatr Clin N Am. 2008 Oct;17(4):887-905, x-xi. doi: 10.1016/j.chc.2008.06.005. PMID 18775376
- [Background] Ledford JR, Gast DL. Feeding problems in children with autism spectrum disorders: A review. Focus Autism Other Dev Disabl. 2006;21(3):153-166
- [Background] Marquenie K, Rodger S, Mangohig K, Cronin A. Dinnertime and bedtime routines and rituals in families with a young child with an autism spectrum disorder. Aust Occup Ther J. 2011 Jun;58(3):145-54. doi: 10.1111/j.1440-1630.2010.00896.x. Epub 2011 Jan 9. PMID 21599679
- [Background] Sharp WG, Berry RC, McCracken C, Nuhu NN, Marvel E, Saulnier CA, Klin A, Jones W, Jaquess DL. Feeding problems and nutrient intake in children with autism spectrum disorders: a meta-analysis and comprehensive review of the literature. J Autism Dev Disord. 2013 Sep;43(9):2159-73. doi: 10.1007/s10803-013-1771-5. PMID 23371510
- [Background] Kral TV, Eriksen WT, Souders MC, Pinto-Martin JA. Eating behaviors, diet quality, and gastrointestinal symptoms in children with autism spectrum disorders: a brief review. J Pediatr Nurs. 2013 Nov-Dec;28(6):548-56. doi: 10.1016/j.pedn.2013.01.008. Epub 2013 Mar 24. PMID 23531467
- [Background] Estes A, Munson J, Dawson G, Koehler E, Zhou XH, Abbott R. Parenting stress and psychological functioning among mothers of preschool children with autism and developmental delay. Autism. 2009 Jul;13(4):375-87. doi: 10.1177/1362361309105658. PMID 19535467
- [Background] Lovell B, Moss M, Wetherell MA. The psychophysiological and health corollaries of child problem behaviours in caregivers of children with autism and ADHD. J Intellect Disabil Res. 2015 Feb;59(2):150-7. doi: 10.1111/jir.12081. Epub 2013 Jul 24. PMID 23889770
- [Background] Dawson G, Rogers S, Munson J, Smith M, Winter J, Greenson J, Donaldson A, Varley J. Randomized, controlled trial of an intervention for toddlers with autism: the Early Start Denver Model. Pediatrics. 2010 Jan;125(1):e17-23. doi: 10.1542/peds.2009-0958. Epub 2009 Nov 30. PMID 19948568
- [Background] Hardan AY, Gengoux GW, Berquist KL, Libove RA, Ardel CM, Phillips J, Frazier TW, Minjarez MB. A randomized controlled trial of Pivotal Response Treatment Group for parents of children with autism. J Child Psychol Psychiatry. 2015 Aug;56(8):884-92. doi: 10.1111/jcpp.12354. Epub 2014 Oct 27. PMID 25346345
- [Background] Rogers SJ, Estes A, Lord C, Vismara L, Winter J, Fitzpatrick A, Guo M, Dawson G. Effects of a brief Early Start Denver model (ESDM)-based parent intervention on toddlers at risk for autism spectrum disorders: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2012 Oct;51(10):1052-65. doi: 10.1016/j.jaac.2012.08.003. Epub 2012 Aug 28. PMID 23021480
- [Background] Manikam R, Perman JA. Pediatric feeding disorders. J Clin Gastroenterol. 2000 Jan;30(1):34-46. doi: 10.1097/00004836-200001000-00007. PMID 10636208
- [Background] Winston KA, Dunbar SB, Reed CN, Francis-Connolly E. Mothering occupations when parenting children with feeding concerns: a mixed methods study. Can J Occup Ther. 2010 Jun;77(3):181-9. doi: 10.2182/cjot.2010.77.3.8. PMID 20597379
- [Background] Ahearn WH, Castine T, Nault K, Green G. An assessment of food acceptance in children with autism or pervasive developmental disorder-not otherwise specified. J Autism Dev Disord. 2001 Oct;31(5):505-11. doi: 10.1023/a:1012221026124. PMID 11794415
- [Background] Martins Y, Young RL, Robson DC. Feeding and eating behaviors in children with autism and typically developing children. J Autism Dev Disord. 2008 Nov;38(10):1878-87. doi: 10.1007/s10803-008-0583-5. Epub 2008 May 16. PMID 18483843
- [Background] Schreck KA, Williams K, Smith AF. A comparison of eating behaviors between children with and without autism. J Autism Dev Disord. 2004 Aug;34(4):433-8. doi: 10.1023/b:jadd.0000037419.78531.86. PMID 15449518
- [Background] Nadon G, Feldman DE, Dunn W, Gisel E. Mealtime problems in children with autism spectrum disorder and their typically developing siblings: a comparison study. Autism. 2011 Jan;15(1):98-113. doi: 10.1177/1362361309348943. Epub 2010 May 18. PMID 20484003
- [Background] Provost B, Crowe TK, Osbourn PL, McClain C, Skipper BJ. Mealtime behaviors of preschool children: comparison of children with autism spectrum disorder and children with typical development. Phys Occup Ther Pediatr. 2010 Aug;30(3):220-33. doi: 10.3109/01942631003757669. PMID 20608859
- [Background] Dabrowska A, Pisula E. Parenting stress and coping styles in mothers and fathers of pre-school children with autism and Down syndrome. J Intellect Disabil Res. 2010 Mar;54(3):266-80. doi: 10.1111/j.1365-2788.2010.01258.x. Epub 2010 Feb 8. PMID 20146741
- [Background] Lecavalier L, Leone S, Wiltz J. The impact of behaviour problems on caregiver stress in young people with autism spectrum disorders. J Intellect Disabil Res. 2006 Mar;50(Pt 3):172-83. doi: 10.1111/j.1365-2788.2005.00732.x. PMID 16430729
- [Background] Greer AJ, Gulotta CS, Masler EA, Laud RB. Caregiver stress and outcomes of children with pediatric feeding disorders treated in an intensive interdisciplinary program. J Pediatr Psychol. 2008 Jul;33(6):612-20. doi: 10.1093/jpepsy/jsm116. Epub 2007 Dec 3. PMID 18056140
- [Background] Laud RB, Girolami PA, Boscoe JH, Gulotta CS. Treatment outcomes for severe feeding problems in children with autism spectrum disorder. Behav Modif. 2009 Sep;33(5):520-36. doi: 10.1177/0145445509346729. Epub 2009 Sep 10. PMID 19748900
- [Background] Baranek GT, Watson LR, Turner-Brown L, Field SH, Crais ER, Wakeford L, Little LM, Reznick JS. Preliminary efficacy of adapted responsive teaching for infants at risk of autism spectrum disorder in a community sample. Autism Res Treat. 2015;2015:386951. doi: 10.1155/2015/386951. Epub 2015 Jan 11. PMID 25648749
- [Background] Bandini LG, Anderson SE, Curtin C, Cermak S, Evans EW, Scampini R, Maslin M, Must A. Food selectivity in children with autism spectrum disorders and typically developing children. J Pediatr. 2010 Aug;157(2):259-64. doi: 10.1016/j.jpeds.2010.02.013. Epub 2010 Apr 1. PMID 20362301
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Boyd BA, McDonough SG, Rupp B, Khan F, Bodfish JW. Effects of a family-implemented treatment on the repetitive behaviors of children with autism. J Autism Dev Disord. 2011 Oct;41(10):1330-41. doi: 10.1007/s10803-010-1156-y. PMID 21161576
- [Background] Pfeiffer B, Kinnealey M. Treatment of sensory defensiveness in adults. Occup Ther Int. 2003;10(3):175-84. doi: 10.1002/oti.184. PMID 12900790
- [Background] Schaaf R, Blanche EI. Comparison of behavioral intervention and sensory-integration therapy in the treatment of challenging behavior. J Autism Dev Disord. 2011 Oct;41(10):1436-8; author reply 1439-41. doi: 10.1007/s10803-011-1303-0. No abstract available. PMID 21667199
- [Background] Ruble L, McGrew JH, Toland MD. Goal attainment scaling as an outcome measure in randomized controlled trials of psychosocial interventions in autism. J Autism Dev Disord. 2012 Sep;42(9):1974-83. doi: 10.1007/s10803-012-1446-7. PMID 22271197
- [Background] Crawford PB, Obarzanek E, Morrison J, Sabry ZI. Comparative advantage of 3-day food records over 24-hour recall and 5-day food frequency validated by observation of 9- and 10-year-old girls. J Am Diet Assoc. 1994 Jun;94(6):626-30. doi: 10.1016/0002-8223(94)90158-9. PMID 8195550
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405